CLINICAL TRIAL: NCT03585335
Title: Development of a Cardiorespiratory Risk Surveillance Score Via Comparison of Body Composition Methods, Cardiorespiratory Fitness, and Obesity in Firefighters
Brief Title: Firefighter Cardiorespiratory Fitness (CRF) Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Due to COVID-19 restrictions and the closure of the research clinic site, the study ended prematurely. Not all data was collected on all participants.
Sponsor: HealthPartners Institute (Other)
Collaborators: Hologic, Inc. (Industry); Performance Plus, LLC (DBA Health Strategies) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IIT-17-01
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2020-12

CONDITIONS: Cardiorespiratory Fitness
Keywords: Cardiorespiratory Fitness Score; BMI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiorespiratory fitness is of vital importance to firefighters and yet is rarely, if ever, tested in a systematic fashion over the course of an individual firefighter's career. Investigators know that there are incremental health benefits to increased levels of fitness and reduced morbidity and mortality associated with lower levels of fitness. The proposed study will address this gap by enrolling up to 135 firefighters from local metropolitan fire departments. The goal of this cross-sectional correlational study is to address which body composition methods best correlate with cardiorespiratory fitness (CRF) in firefighters in order to define a method to combine data into a risk score predictive of fitness. Specifically, this study will 1) measure body composition data and evaluate the correlation of BMI with non-BMI body composition measures, such as body fat percentage (BF%), lean body mass percentage (LBM%), or waist circumference (WC), 2) measure cardiorespiratory fitness in terms of VO2max and evaluate the correlation of body composition measures such as BMI, BF%, LBM%, and/or WC with VO2max,, 3) evaluate diagnostic test metrics, such as sensitivity and specificity, of population meeting obesity criteria by BMI and WC, as compared to BF% as the reference standard, 4) develop a cardiorespiratory fitnessscore (CVFS) from a conjunction of body composition measures (BMI, as BF%, LBM%, WC) and demographic variables that is well-correlated with measured VO2max, evaluate the CVFS performance in age and gender-stratified subpopulations relative to the accepted standard of gender-stratified VO2max criteria, and identify age and gender-stratified CVFS threshold and diagnostic test performance; and 5) correlate CVFS performance with cardiovascular risk measures. Results of this analysis will provide pilot data and inform future work to assess whether providing more accurate data on body composition can lead to more effective reductions in cardiorespiratory risk in this population.

DETAILED DESCRIPTION:
Firefighters are exposed to extreme metabolic and cardiopulmonary stressors in the performance of their vocation that are recognized to exceed the actual physical or environmental hazards. The current medical literature regarding firefighting highlights two frequently cited statistics: (1) based on body mass index (BMI), upwards of 73-80% of firefighters are considered overweight or obese, and (2) >45% of firefighter line-of-duty deaths are due to cardiovascular events.

This finding regarding BMI has been widely reported in the U.S. media after being published in a 2014 CDC medical journal. Such a finding is particularly relevant to firefighters given that there are recommended cardiorespiratory performance standards for firefighters, commonly 12 metabolic equivalents (METs) or maximum oxygen consumption during aerobic exercise (VO2max) of 42 mL O2/kg of body weight/min. As a consequence, failure to meet such a standard may limit a firefighter's ability to perform (or be employed) in full-duty tasks based on individual fire station requirements.

Fire suppression activities account for 1-5% of a firefighter's duty time yet result in 32% of firefighter deaths. This is attributable to the extreme physical demands of firefighting activities in which anaerobic threshold (typically 85% of maximal heart rate) may be exceeded and sustained throughout an engagement. Few professions, other than elite athletes, require this level of cardiorespiratory fitness (CRF). As such, CRF is of vital importance to firefighters and yet is rarely, if ever, tested in a systematic fashion over the course of an individual firefighter's career.

The vital importance of CRF is well-established in the medical literature, such that many advocate for its addition as a clinical vital sign. Epidemiological studies have demonstrated an inverse relationship between CRF and coronary heart disease (CHD) and all-cause mortality in healthy individuals. There are incremental health benefits to increased levels of fitness and reduced morbidity and mortality associated with lower levels of fitness. The fitness standard of 12 METs (the equivalent of a VO2max of 42 mL/kg/min) remains the testing metric for firefighters in the NFPA 1582 guidelines; it is applied to all candidates, male or female, and of any age. While a VO2max of 42 may be "good" to "excellent" for a 50-59 year old male, it is only "good" for a 40-49 year old male, and only "fair" for a 30-39 or "poor" for a 20-29 year old male. In women, a VO2max of 42 indicates a "good" level of CRF for a 20-29 year old female and "superior" CRF for a 50-59 year old female. Knowing that CRF declines inevitably with age argues that a firefighter whose VO2max is 42 mL/kg/min at age 20 will decline significantly by age 50 and raises the question of their ability to safely participate in fire suppression activities at that age. CRF measures in firefighters would benefit from age-adjustment and gender stratification. This research would begin that process.

While elevated BMI is associated with cardiovascular disease morbidity and mortality, BMI has been demonstrated to be a non-specific metric of body composition. Specifically, BMI "is limited as an index of obesity (body fatness) because it does not account for the composition of body weight," and the concurrence of BMI and body fat percentage (BF%) is affected by age, gender, ethnicity, and body shape. The misclassification of firefighters as overweight and obese based on BMI has been discussed in a several studies. These studies utilized bioimpedance testing or skin calipers for BF% measurement, methods known to have significant levels of error in terms of false positives and false negatives. Interestingly, a series of these studies cite a single article with a sample size of 39 individuals as validation of bioimpedance in comparison to dual-energy X-ray absorption (DXA), but also report DXA as the gold standard for BF% measurement. This inaccuracy of BF% compared to BMI was addressed thoroughly in one study of U.S. firefighters, demonstrating the potential for false positive and false negative identification of obesity in this population; specifically, they reported rates of 15.4% false positive and 18.2% false negative identification of obesity when identified by BMI as opposed to BF%.

The primary advantages of using BMI in a clinical setting include the long-established history of BMI usage and its extremely low cost (simply measuring someone's height and weight). However, waist circumference (WC) is easily measured, and has demonstrated comparable prediction of cardiovascular risk as compared to and in conjunction with BMI.10 Although classification of obesity has not been conducted by WC, an elevated cardiovascular risk has been identified for men with WC > 102 cm and women with WC > 88 cm.More specifically, WC classifications of very low, low, high, and very high have been developed. For purposes of this study, WC measurements within the high and very high classifications are considered as obese, with this population (WC > 100 cm in males, WC > 90 cm in females) representing a similar population to those identified with an increased cardiovascular risk.

The knowledge gap between BF% and cardiovascular risk as it pertains to clinical use of BMI and other body composition metrics has been identified by the National Heart, Lung, and Blood Institute (NHLBI), whose 2013 systematic review noted, "studies using BMI and waist circumference compared to more valid measures of percent body fat are needed to examine the predictive role of various adiposity measures." However, strong correlations between body composition metrics and CRF were found in a recent study in Brazilian firefighters, and in this case, BMI was considered to be an adequate surrogate for other body composition methods evaluating body composition. A limitation of this study was that it used skin caliper testing for BF% measurement and a non-respiratory-based exercise test to indirectly estimate VO2max. Thus, there is an evident need to clarify which among several potential measures of body composition best predicts CRF, with firefighters serving as a relevant population for study. To the best of our knowledge, there are no studies that utilize the accepted criterion standard of dual X-ray energy absorption (DXA) scanning coupled with measured VO2max testing that would allow coupling these two metrics into a reference fitness-leanness measure.

DXA is a widely-available technology that is relatively inexpensive compared with other diagnostic technologies, is safe, and can accurately measure BF%. DXA studies can be completed in less than ten minutes and provide data that is valid and reproducible over time. The radiation from a DXA scan is less than that received from routine environmental exposure in a single day. Americans typically receive approximately 3.0 milliSieverts (mSv) of radiation exposure annually from cosmic radiation, household radon, and other environmental sources. This does not include elective diagnostic imaging sources. The radiation exposure of a DXA scan is ~0.005 mSv, about a tenth of that from a single chest x-ray (CXR). 19 By comparison a CT scan of the pelvis, chest or abdomen can expose the patient to 6.0 -10.0 mSv in one study (the equivalent of 2-3 years of environmental exposure in a single medical study). A CT scan of the head is ~2.0 mSv.20 A lumbar spine X-ray series is ~1.5 mSv and a single PA (posterior-anterior) chest X-ray (CXR) is ~0.06 mSv. The precept of As Low As Reasonably Achievable (ALARA) in order to minimize radiation exposure is easily honored in the case of DXA scanning due to the extremely low mSv exposures. The Biological Effects of Ionizing Radiation (BEIR) VII report and executive summary provide definitive recommendations regarding radiation exposure and cancer risk.

DXA has been identified an accurate method of measuring BF%, with the additional benefit of also measuring lean body mass percentage (LBM%) and, of course, bone mineral density (BMD), as well. This is supported by numerous studies including BF% measured by DXA as the reference against their study variable of interest. Obesity has been defined for BF% by age categories, with classifications of low, mid, high, and obesity, where the bottom of the low range is the minimum of essential body fat. On the other hand, LBM% has not been extensively studied in correlation with obesity in adults, though contemporary work has been conducted to estimate LBM% in children and adolescents.

As such, this study aims to address which body composition methods best correlate with CRF in firefighters. Investigators hypothesize that BF% will better correlate with CRF metrics than traditional (but technologically outdated) body composition methods, such as BMI or waist circumference (WC), and furthermore in conjunction with measurement of LBM%. Additionally, investigators hypothesize that these data, in conjunction with demographic, employment, physical activity, and medical history data, can comprise a simplified metric (a cardiorespiratory fitness score) to estimate firefighter CRF. In this context, a cost analysis of the evaluated surveillance methods will be generated.

Cardiovascular risk has been evaluated in the context of CRF previously, but not specifically in terms of correlating VO2max and cardiovascular risk measures in firefighters. Most recently, Yang et al. reported significantly decreased cardiovascular risk in a firefighter population relative to increased number of push-ups performed.24 A well-accepted measure of cardiovascular risk in adults is the Framingham Risk Score, which estimates a percentage of cardiovascular disease risk over 10 years as a function of age, serum cholesterol measures, blood pressure, diabetes history, and smoking status; this tool is often considered the gold standard of evaluating 10-year cardiovascular disease risk.25 Studies have demonstrated an inverse association between CRF - in terms of VO2max or otherwise - and the Framingham Risk Score, in a variety of populations, including men, women, and diabetics.26-30 Notably, Gander et al. (2017) specifically discussed the added utility of correlating Framingham Risk with estimated cardiorespiratory fitness in an asymptomatic male population, which to some degree may mimic much of the firefighter population, wherein most are primarily male and asymptomatic.31 This study aims to add to the literature base demonstrating that higher cardiorespiratory fitness is correlated with lower cardiovascular risk, but uniquely in the context of the firefighter population. As cardiorespiratory fitness is a good measure of performance, the concurrent demonstration of decreased cardiovascular risk in a cost-effective way can add significant value to evaluation of firefighters, in whom these more elevated risks have been identified.

Results of this analysis will provide pilot data and inform future work to assess whether providing more accurate data on body composition can lead to more effective reductions in cardiorespiratory risk in this population. This study has the additional benefit of creating the availability of DXA three-compartment (fat mass, lean mass, bone mineral content) body composition at our institution, where this study is not currently performed despite the required technology already being used for bone studies.

ELIGIBILITY:
Phase I: Inclusion Criteria:

1. Fire fighter from selected local metropolitan fire department(s)
2. Willing and agree to complete all data collection components of the study - Anthropometrics, participant survey, Concept 2 Rower Test 2,000 meter test, Treadmill VO2max Test, and DXA scan

Phase II Inclusion Criteria:

1. Fire fighter from selected local metropolitan fire department(s)
2. Willing and agree to complete all data collection components of the study - Anthropometrics, participant survey, Concept 2 Rower Test 2,000 meter test, Treadmill VO2max Test, and DXA scanDXA scan, and electronic data transmission of annual blood pressure and serum cholesterol surveillance data or collection of blood pressure and serum cholesterol

Phase I and Phase II: Exclusion Criteria:

1. Declined participation in the study
2. Unwilling or do not agree to complete all data collection components of the study
3. Pregnant females or females who anticipate being pregnant during the course of the study due to administration of the VO2max fitness test and DXA scan (pregnancy may not appropriately reflect an active-duty firefighter's cardiorespiratory fitness and radiation exposure will be avoided in pregnant individuals)
4. Those who are not currently authorized to operate at full duty with their fire department without restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 135 firefighters from local metropolitan fire departments will be enrolled in this study. To minimize selection bias, although individual firefighters may opt out of the study, an attempt will be made to enroll all firefighters from an individual department to minimize volunteer bias.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Multivariate prediction score of cardiorespiratory risk | 2 months
  Develop a cardiorespiratory fitness score (CVFS) from a conjunction of body composition measures (Body Mass Index [BMI], as body fat percentage [BF%], lean body mass percentage [LBM%], and waist circumference [WC]) and demographic variables that is well-correlated with measured VO2max, evaluate the cardiorespiratory risk score performance in age and gender-stratified subpopulations relative to the accepted standard of gender-stratified VO2max criteria, and identify age and gender-stratified cardiorespiratory risk score threshold and diagnostic test performance.

SECONDARY OUTCOMES:
Correlation of non-body mass index (BMI) body composition methods with body mass index | 2 months
  Measure body composition data and evaluate the correlation of body mass index (BMI) with non-body mass index body composition measures, such as body fat percentage (BF%), lean body mass percentage (LBM%), or waist circumference (WC) in individuals in a firefighter population.
Correlation of body composition methods with measured VO2max | 2 months
  Measure cardiorespiratory fitness in terms VO2max and evaluate the correlation of body composition measures such as body mass index (BMI), body fat percentage (BF%), lean body mass percentage (LBM%), and/or waist circumference (WC) with VO2max, in individuals in a firefighter population.
Diagnostic test evaluation of body composition methods for meeting obesity criteria | 2 months
  Evaluate diagnostic test metrics, such as sensitivity and specificity, of population meeting obesity criteria by body mass index (BMI) and waist circumference (WC), as compared to body fat percentage (BF%) as the reference standard.
Direct estimated cost comparison of measured VO2max with developed prediction score | 2 months
  Estimate cost-effectiveness of a developed cardiorespiratory risk score in comparison to measured VO2max in a firefighter population.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States